CLINICAL TRIAL: NCT02354352
Title: Therapeutic Potential for Aldosterone Inhibition in Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of California, Los Angeles (Other); University of Utah (Other); University of Colorado, Denver (Other); University of Kansas Medical Center (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Subha Raman, Professor of Medicine, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014H0387
Record Dates: First submitted 2015-01-27; First posted 2015-02-03 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Eplerenone; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eplerenone (Active Comparator): Eplerenone is an aldosterone antagonist used as an adjunct in the management of chronic heart failure. It is marketed under the trade name Inspra. Eplerenone is a potassium-sparing diuretic.
  Interventions: Drug: Eplerenone
- Spironolactone (Active Comparator): Spironolactone is an aldosterone antagonist used as an adjunct in the management of chronic heart failure. It is marketed under the trade name Aldactone. Spironolactone is a potassium-sparing diuretic.
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Eplerenone — 26 Subjects will take Eplerenone, one 50mg capsule by mouth once daily for 12 months.
  Other Names: Inspra
  Arms: Eplerenone
Drug: Spironolactone — 26 Subjects will take Spironolactone, one 50mg capsule by mouth once daily for 12 months.
  Other Names: Aldactone
  Arms: Spironolactone

SUMMARY:
The study is to demonstrate non-inferiority of spironolactone vs. eplerenone in preserving cardiac and pulmonary function in patients with preserved LV ejection fraction. Males with Duchenne muscular dystrophy (DMD) confirmed clinically and by mutation analysis will be enrolled. Subjects will be randomized to either eplerenone or spironolactone. Subjects will use a drug diary to record daily compliance of taking the study medication as well as any concerns they may have during the study period. Subjects will undergo cardiac magnetic resonance imaging (CMR) and pulmonary function tests (PFT) at baseline and then again at 12 months post enrollment. Subjects will also complete a quality of life questionnaire at baseline and 12 months. Degree of elbow contracture will be measured using a goniometer at baseline and 12 months.

DETAILED DESCRIPTION:
DMD is an X-linked disorder in which the sarcolemmal protein dystrophin is effectively absent. Males with DMD typically die in the third and fourth decades of life of cardiopulmonary disease. Mouse models of DMD, autopsy data, and in vivo human studies using magnetic resonance-based late gadolinium enhancement imaging (LGE) have shown that progressive myocardial damage is well underway before left ventricular ejection fraction (LV EF) becomes abnormal.

Exertional symptoms and signs of myocardial disease are typically absent as skeletal muscle disease progressively limits functional capacity in affected boys. Thus, cardiac involvement can go undetected until LV dysfunction and myocardial fibrosis are advanced. While echocardiography remains a useful tool to evaluate LV dysfunction, CMR with LGE is advantageous for DMD patients since it identifies myocardial injury before decline in EF is apparent by echocardiography. Further, greater reproducibility affords efficient sample sizes for cardiomyopathy clinical trials in patients with rare diseases. CMR's increasing availability at DMD clinical centers has afforded earlier cardiomyopathy detection, and has helped refine current management to typically include agents such as angiotensin converting enzyme inhibitors (ACEI) once damage is evident. This strategy, however, may not be sufficient, with prior studies showing decline in systolic function with or without ACEI or angiotensin receptor blocker (ARB) therapy.

The investigators previously tested mineralocorticoid receptor antagonism (MRA) added to ACEI while EF was still normal in a mouse model that mimics the myocardial damage seen in DMD patients. This combination significantly reduced myocardial injury and improved (made more negative) LV circumferential strain (Ecc), a sensitive and early marker of LV systolic dysfunction. Additionally, preliminary findings from a recently completed clinical trial suggests efficacy of eplerenone vs. placebo, while further preclinical data suggests greater benefit without concomitant steroid use. Thus, a non-inferiority trial comparing MRAs is needed.

ELIGIBILITY:
Inclusion Criteria:

* Boys age ≥7 years with DMD confirmed clinically and by mutation analysis able to undergo cardiac magnetic resonance (CMR) without sedation
* LV EF ≥45% (+/-5%) by clinically-acquired echocardiography, nuclear scan or cardiac MRI done within 2 weeks of enrollment

Exclusion Criteria:

* Non-MR compatible implants
* Severe claustrophobia
* Gadolinium contrast allergy
* Kidney disease
* Prior use of or allergy to aldosterone antagonist
* Use of other investigational therapy.

Min Age: 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subha V Raman, MD, Principal Investigator — Ohio State University
Locations (6):
- United States (6):
  - Mattel Children's Hospital and David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - University of Kansas Medical Center, Kansas City, Kansas
  - The Ohio State University Medical Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raman SV, Hor KN, Mazur W, Cardona A, He X, Halnon N, Markham L, Soslow JH, Puchalski MD, Auerbach SR, Truong U, Smart S, McCarthy B, Saeed IM, Statland JM, Kissel JT, Cripe LH. Stabilization of Early Duchenne Cardiomyopathy With Aldosterone Inhibition: Results of the Multicenter AIDMD Trial. J Am Heart Assoc. 2019 Oct;8(19):e013501. doi: 10.1161/JAHA.119.013501. Epub 2019 Sep 24. PMID 31549577

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eplerenone | Spironolactone
Started | 26 | 26
2 Weeks | 26 | 25
1 Month | 24 | 23
2 Months | 24 | 22
3 Months | 25 | 23
6 Months | 25 | 23
9 Months | 25 | 23
Completed | 23 | 23
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eplerenone | Spironolactone | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 19 | 40
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14 [13 to 18] | 13 [12 to 20] | 14 [12 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 26 | 26 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 24 | 20 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 24 | 25 | 49
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Ambulatory [Count of Participants; unit: Participants] | 4 | 6 | 10
Nocturnal ventilatory support [Count of Participants; unit: Participants] | 7 | 6 | 13
Forced vital capacity [Mean (Standard Deviation); unit: Liters] — Population: One patient did not receive a pulmonary function test at baseline.
  Liters
    number analyzed (Participants) | 26 | 25 | 51
    (all) | 1.7 (0.8) | 1.9 (0.8) | 1.8 (0.8)
Dystrophin mutation type [Count of Participants; unit: Participants]
  Exon deletion | 16 | 15 | 31
  Exon duplication | 4 | 3 | 7
  Other | 6 | 8 | 14
Left ventricular ejection fraction [Mean (Standard Deviation); unit: Percent of blood ejected from LV] — Population: One patient did not have adequate MRI images for analysis of this measure.
  Percent of blood ejected from LV
    number analyzed (Participants) | 26 | 25 | 51
    (all) | 55 (8.7) | 57 (7.6) | 56 (8.2)
Left ventricular circumferential strain [Mean (Standard Deviation); unit: Percent change in circumference] — Population: One patient did not have adequate MRI images for analysis of this measure.
  Percent change in circumference
    number analyzed (Participants) | 25 | 26 | 51
    (all) | -14.5 (2.70) | -14.2 (2.16) | -14.3 (2.42)
Late gadolinium enhancement [Mean (Standard Deviation); unit: Percent of enhanced myocardium] — Population: Several patients did not have adequate MRI images for analysis of this measure.
  Percent of enhanced myocardium
    number analyzed (Participants) | 22 | 24 | 46
    (all) | 10.3 (10.7) | 14.5 (14.7) | 12.5 (12.9)
Blood pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 112.6 (14.1) | 118.5 (14.7) | 115.6 (14.6)
  Diastolic | 69.4 (15.7) | 70.8 (11.5) | 70.1 (13.7)
Heart rate [Mean (Standard Deviation); unit: beats per minute] — Population: One patient did not get a heart rate taken at baseline.
  beats per minute
    number analyzed (Participants) | 26 | 25 | 51
    (all) | 95.3 (14.3) | 99.9 (11.9) | 97.5 (13.2)
Weight [Mean (Standard Deviation); unit: kilograms] | 55.6 (15.1) | 55.8 (20.9) | 55.7 (18.1)
Serum potassium [Mean (Standard Deviation); unit: mmol/L] | 4.1 (0.45) | 4.1 (0.50) | 4.1 (0.47)
Background medical therapy [Count of Participants; unit: Participants]
  ACEI | 15 | 15 | 30
  ARB | 2 | 0 | 2
  Beta-blocker | 3 | 7 | 10
  Any Steroid Use, Current or Previous | 21 | 23 | 44
  Prednisone | 15 | 11 | 26
  Deflazacort | 6 | 12 | 18

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Strain
Description: a sensitive measure of heart muscle function
Time Frame: 12 months
Population: One patient in the spironolactone group did not receive a follow-up MRI.
Measure: Median (Inter-Quartile Range); unit: Percent change in circumference
Arm/Group | Eplerenone | Spironolactone
Number analyzed (Participants) | 23 | 22
Percent change in circumference | 0.2 [-0.2 to 0.7] | 0.4 [-0.4 to 1.0]
Statistical Analysis 1: Comparison: Eplerenone vs Spironolactone; Test type: Non-Inferiority — Using a Type I error rate of 5%, we conducted a power calculation using a non-inferiority test on 12-month change in Ecc. If there is truly no difference in the 12-month Ecc change between the spironolactone and eplerenone groups, 46 patients (23 in each group) would result in at least 80% power to ensure that the lower limit of a one-sided 95% confidence interval for the true difference between the spironolactone and eplerenone groups to be above the non-inferiority limit of -1.75; p = 0.5867, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Description: The definitions used to collect adverse event information did not differ from the clinicaltrials.gov definitions.
Arm/Group | Eplerenone | Spironolactone
All-Cause Mortality (participants affected / at risk) | 2/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 3/26 | 2/26
Other Adverse Events (participants affected / at risk) | 2/26 | 3/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eplerenone (N=26) | Spironolactone (N=26)
Accidental Drowning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Participant was found face down in irrigation canal after experimenting with LSD.
Pneumonia Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) — Requiring hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eplerenone (N=26) | Spironolactone (N=26)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gynecomastia (Endocrine disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT02354352/Prot_SAP_000.pdf